CLINICAL TRIAL: NCT00803998
Title: Ocular Hypertension Treatment Study
Brief Title: Ocular Hypertension Treatment Study (OHTS)
Status: Completed | Type: Observational
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Other Study IDs: 93.01
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2008-12

CONDITIONS: Ocular Hypertension; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

SUMMARY:
The Ocular Hypertension Treatment Study is a multi-center clinical trial sponsored by the National Eye Institute, designed to determine the efficacy and safety of topically administered eye lowering medication

ELIGIBILITY:
Inclusion Criteria:

* Qualifying IOP in at least one eye of each participant must be more than or equal 24 mmHg but less than or equal to 32 mm HG calculated from two separate consecutive determination taken at least 2 hours, but not greater than 12 weeks apart.
* Normal and reliable 30-2 Humphrey Visual Fields in both eyes.
* Normal Optic disc in both eyes on clinical examinations and stereoscopic photographs as determined by the Optic Disc Reading Center.

Exclusion Criteria:

* Visual acuity worse than 20/40 in either eye on qualifying exam.
* Previous intraocular surgery: laser trabeculoplasty, laser iridotomy, filtering surgery, combined cataract extraction/filtering procedures, penetrating keratoplasty and retinal detachment repair.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1994-02; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kass, MD, Study Chair — Washington University School of Medicine at St. Louis, St. Louis, Missouri

REFERENCES:
- [Background] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575